CLINICAL TRIAL: NCT02796573
Title: Blended Cognitive Behavioural Therapy Versus Face-to-face Cognitive Behavioural Therapy: A Randomised Non-inferiority Trial
Brief Title: Blended Cognitive Behavioural Therapy Versus Face-to-face Cognitive Behavioural Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kim Mathiasen, Ph.D. fellow, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20150150
Record Dates: First submitted 2016-06-01; First posted 2016-06-10 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Adult Depression
Keywords: blended care; CBT; B-CBT; depression
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- B-CBT (Experimental): 6 face-to-face consultations plus 6 online modules.
  Interventions: Behavioral: cognitive behavioural therapy
- Face-to-Face CBT (Active Comparator): 12 face-to-face consultations.
  Interventions: Behavioral: cognitive behavioural therapy

INTERVENTIONS:
Behavioral: cognitive behavioural therapy

SUMMARY:
Depression is a prevalent and disabling disorder with great cost to the individual and the society. Lately, the use of internet interventions as guided self-help has demonstrated remarkable results. However, certain shortcomings such as lack of personal adaptation has been identified.

The presents study aims to investigate the potential of blending Internet based interventions with face-to-face consultations using cognitive behavioural therapy (B-CBT). The main hypotheses are, that that B-CBT will be as clinically effective as TAU, and that it will be acceptable to patients and clinicians.

The study is designed as a two arm randomised non-inferiority trial comparing internet based B-CBT for depression to treatment as usual (TAU) defined as 12 sessions of face-to-face CBT.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older.
* Meet Diagnostic and Statistic Manual of Mental Disorders 4th. edition (DSM-IV) diagnostic criteria for major depressive disorder as confirmed by the telephone administered Mini International Neuropsychiatric Interview version 5.0 (MINI)and a score of 5 or higher on the Patient Health Questionnaire nine items (PHQ-9).

Exclusion Criteria:

* Current high risk of suicide according to the MINI Interview section C.
* Co-morbid substance dependence, bipolar affective disorder, psychotic illness, obsessive compulsive disorder, as established at the MINI interview.
* Currently receiving psychological treatment for depression in primary or specialised mental health care
* Being unable to comprehend the spoken and written language of Danish.
* Not having access to a computer and fast Internet connection (i.e. broadband or comparable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-03; Primary Completion 2019-05-01 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9-item change | Change from Baseline, 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Telepsychiatry, Odense, Fyn, Denmark

REFERENCES:
- [Derived] Doukani A, Quartagno M, Sera F, Free C, Kakuma R, Riper H, Kleiboer A, Cerga-Pashoja A, van Schaik A, Botella C, Berger T, Chevreul K, Matynia M, Krieger T, Hazo JB, Draisma S, Titzler I, Topooco N, Mathiasen K, Vernmark K, Urech A, Maj A, Andersson G, Berking M, Banos RM, Araya R. Comparison of the Working Alliance in Blended Cognitive Behavioral Therapy and Treatment as Usual for Depression in Europe: Secondary Data Analysis of the E-COMPARED Randomized Controlled Trial. J Med Internet Res. 2024 May 31;26:e47515. doi: 10.2196/47515. PMID 38819882
- [Derived] Mathiasen K, Andersen TE, Lichtenstein MB, Ehlers LH, Riper H, Kleiboer A, Roessler KK. The Clinical Effectiveness of Blended Cognitive Behavioral Therapy Compared With Face-to-Face Cognitive Behavioral Therapy for Adult Depression: Randomized Controlled Noninferiority Trial. J Med Internet Res. 2022 Sep 7;24(9):e36577. doi: 10.2196/36577. PMID 36069798
- [Derived] Mathiasen K, Andersen TE, Riper H, Kleiboer AA, Roessler KK. Blended CBT versus face-to-face CBT: a randomised non-inferiority trial. BMC Psychiatry. 2016 Dec 5;16(1):432. doi: 10.1186/s12888-016-1140-y. PMID 27919234